CLINICAL TRIAL: NCT02967380
Title: Dynamic Contrast Enhanced Steady State T1-Weighted Perfusion MRI (DCE MRI): Characterization of Intracranial Lesions
Brief Title: Gadobutrol Versus Gadopentetate Dimeglumine or Gadobenate Dimeglumine Before DCE-MRI in Diagnosing Patients With Multiple Sclerosis, Grade II-IV Glioma, or Brain Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient Accrual
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0S-11-6; NCI-2014-01852 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); D1 2010-10; HS-11-00363; 0S-11-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-09-13; First posted 2016-11-18 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Adult Anaplastic (Malignant) Meningioma; Adult Anaplastic Astrocytoma; Adult Anaplastic Ependymoma; Adult Anaplastic Oligodendroglioma; Adult Brain Stem Glioma; Adult Choroid Plexus Neoplasm; Adult Diffuse Astrocytoma; Adult Ependymoblastoma; Adult Ependymoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Grade II Meningioma; Adult Medulloblastoma; Adult Mixed Glioma; Adult Oligodendroglioma; Adult Papillary Meningioma; Adult Pineal Gland Astrocytoma; Adult Pineoblastoma; Adult Primary Melanocytic Lesion of Meninges; Adult Supratentorial Primitive Neuroectodermal Tumor; Malignant Adult Intracranial Hemangiopericytoma; Metastatic Malignant Neoplasm in the Brain; Multiple Sclerosis; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Meningioma; Astrocytoma; Ependymoma; Oligodendroglioma; Choroid Plexus Neoplasms; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Glioma; Pinealoma; Brain Neoplasms; Multiple Sclerosis | interventions — gadobenic acid; gadobutrol; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Magnevist/Multihance, Gadavist, DCE-MRI) (Experimental): Patients receive standard of care gadopentetate dimeglumine IV twice within 5 minutes or gadobenate dimeglumine IV twice within 5 minutes and then undergo DCE-MRI on day 1. Patients also receive gadobutrol IV twice within 5 minutes and then undergo DCE-MRI over approximately 30 minutes on day 3, 4, 5, 6, or 7.
  Interventions: Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging; Drug: Gadobenate Dimeglumine; Drug: Gadobutrol; Radiation: Gadopentetate Dimeglumine

INTERVENTIONS:
Procedure: Dynamic Contrast-Enhanced Magnetic Resonance Imaging — Undergo DCE-MRI
  Other Names: DCE MRI; DCE-MRI; DYNAMIC CONTRAST ENHANCED MRI
Drug: Gadobenate Dimeglumine — Given IV
  Other Names: Gd-BOPTA; MultiHance
Drug: Gadobutrol — Given IV
  Other Names: BAY86-4875; Gadograf; Gadovist; Protovis; ZK 135079
Radiation: Gadopentetate Dimeglumine — Given IV
  Other Names: Gadolinium DTPA; Gd-DTPA; Magnevist; Meglumine Gadopentetate; SH L 451 A; ZK 93035

SUMMARY:
This pilot clinical trial compares gadobutrol with standard of care contrast agents, gadopentetate dimeglumine or gadobenate dimeglumine, before dynamic contrast-enhanced (DCE)-magnetic resonance imaging (MRI) in diagnosing patients with multiple sclerosis, grade II-IV glioma, or tumors that have spread to the brain. Gadobutrol is a type of contrast agent that may increase DCE-MRI sensitivity for the detection of tumors or other diseases of the central nervous system. It is not yet known whether gadobutrol is more effective than standard of care contrast agents before DCE-MRI in diagnosing patients with multiple sclerosis, grade II-IV glioma, or tumors that have spread to the brain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether Gadavist® (gadobutrol) is consistent with Magnevist® (gadopentetate dimeglumine) or Multihance (gadobenate dimeglumine) in the preoperative grading of gliomas utilizing DCE MRI.

II. To determine whether Gadavist® is consistent with Magnevist® or Multihance in identifying the number of cerebral metastases from a primary cancer elsewhere in the body using T1-weighted post contrast MRI.

III. To determine if Gadavist® is consistent with Magnevist® or Multihance in identifying multiple sclerosis (MS) plaques using T1-weighted post contrast MRI.

IV. To determine if Gadavist® produces similar MR perfusion/permeability values of MS lesions as Magnevist® or Multihance.

V. Descriptive analysis to present the different rating patterns of Gadavist® versus Magnevist® or Multihance in differentiating therapeutic necrosis from recurrent tumor in gliomas utilizing DCE MRI.

OUTLINE:

Patients receive standard of care gadopentetate dimeglumine intravenously (IV) twice within 5 minutes or gadobenate dimeglumine IV twice within 5 minutes and then undergo DCE-MRI on day 1. Patients also receive gadobutrol IV twice within 5 minutes and then undergo DCE-MRI over approximately 30 minutes on day 3, 4, 5, 6, or 7.

After completion of study, patients are followed up at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of multiple sclerosis, known or suspected diagnosis of glioma, or known or suspected diagnosis of cerebral metastasis
* Scheduled or to be scheduled for a follow-up MRI per standard of care for their disease
* Minimum permitted time intervals from prior treatments are 6 weeks for intracranial surgery
* Adequate renal function (serum creatinine =< 1.5 mg/dL)
* Subject must sign a study-specific informed consent

Exclusion Criteria:

* Medically unstable
* Renal impairment (glomerular filtration rate [GFR] < 60 mL/min/1.73m^2) or history of existing nephrogenic systemic fibrosis (NSF)
* Cardiac pacemaker
* A serious concurrent infection, illness, or medical condition
* Subjects with any surgical clip, external clips, or any other ferromagnetic device, that is contraindicated for use in MRI
* Subject is claustrophobic and cannot cooperate for the MRI
* Females who are pregnant or nursing
* Any other condition that would compromise the scan with reasonable safety

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12-14 (Actual); Primary Completion 2014-10-14 (Actual); Study Completion 2015-10-14 (Actual)

PRIMARY OUTCOMES:
Agreement of using Magnevist® or Multihance versus Gadavist® on glioma grading | Up to 7 days
  Weighted Kappa analysis will be used to examine the agreement of using Magnevist® or Multihance versus Gadavist® on glioma grading.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Law, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States